CLINICAL TRIAL: NCT04550039
Title: Comparison of Two High-intensity Gait Training Interventions on Contraversive Pushing Behaviors in Individuals Poststroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00213155
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Stroke; Gait; Exoskeleton; Robotics; Contraversive pushing behaviors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Body-weight-supported treadmill training (Experimental): Participants complete prescribed gait training program for at least three weeks or until they discharge.
  Interventions: Device: Body-weight-supported treadmill
- EksoNR exoskeleton (Experimental): Participants complete prescribed gait training program for at least three weeks or until they discharge.
  Interventions: Device: Ekso Bionics EksoNR exoskeleton

INTERVENTIONS:
Device: Body-weight-supported treadmill — Gait training performed on treadmill with overhead harness providing necessary body-weight-support with assistance from trained physical therapist
  Arms: Body-weight-supported treadmill training
Device: Ekso Bionics EksoNR exoskeleton — Gait training performed overground in EksoNR exoskeleton with assistance from trained physical therapist
  Arms: EksoNR exoskeleton

SUMMARY:
The purpose of this study is to investigate the effect of two high-intensity gait training interventions on contraversive pushing behaviors in individuals poststroke in the acute inpatient rehabilitation setting. We will also evaluate the effect of these interventions on functional mobility, strength, balance, and endurance. Furthermore, we intend to measure therapist burden when mobilizing individuals with contraversive pushing behaviors.

DETAILED DESCRIPTION:
High-intensity gait training is strongly supported in individuals poststroke to facilitate neuroplastic changes in the brain in order to maximize the recovery of functional independence. Individuals with contraversive pushing behaviors (CPB) poststroke are difficult to mobilize as a result of tilted posture with significant balance impairments, a tendency to push toward their hemiparetic side, and resistance to external correction. CPB has been reported in 12-18% of individuals receiving stroke rehabilitation and often leads to longer lengths of stay, poorer functional outcomes, and institutionalized discharge locations compared to individuals poststroke without CPB.

High quality evidence guiding physical therapy intervention, specifically gait training, in individuals with CPB is scarce. Traditional therapeutic interventions in individuals with CPB consists of progressing functional mobility while orienting to midline with various forms of visual and tactile feedback. To further guide best practice in this population, we plan to investigate the effect of two high-intensity gait training interventions on CPB in 10 individuals poststroke in the acute inpatient rehabilitation setting over the course of one year.

Individuals from the inpatient stroke unit at the Shirley Ryan AbilityLab will be recruited and placed into one of two intervention groups. Intervention for group one will consist of body-weight-supported treadmill training + overground gait training. Intervention for group two will consist of gait training in the EksoNR exoskeleton + overground gait training. The commercially available EksoNR is approved by the FDA for use in individuals with stroke diagnoses. We will also evaluate the effect of these interventions on functional outcomes including mobility, strength, balance, walking speed, and walking endurance in addition to measuring therapist burden when mobilizing individuals with CPB.

Both groups will receive their specified gait training intervention three sessions a week for at least three weeks until they discharge with the goal of maximizing the number of steps within a 60 minute session. Gait training interventions will be progressed to challenge individuals as appropriate in order to reach 70-85% of age-predicted maximum heart rate. A fourth session will be utilized to assess weekly outcome measures as part of the standard of care at the Shirley Ryan AbilityLab. There will be no restrictions set on therapy delivered outside of these intervention training sessions as individuals will be getting other therapies each day as the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Unilateral, supratentorial ischemic or hemorrhagic stroke within the past six months
* Medical clearance from primary medical team (signed Medical Clearance form)
* Contraversive pushing behaviors as determined by a score of >0 on the Scale for Contraversive Pushing
* Adequate cognitive function as determined by the NIH scale: score ≤1 on question 1b and score =0 on question 1c
* Informed consent provided by participant or power of attorney
* English speaking

Exclusion Criteria:

* Severe aphasia limiting ability to express needs or discomfort verbally or nonverbally
* Severe behavioral neglect as determined by a score of ≥ 21 on Catherine Bergego Scale (CBS) via the Kessler Foundation-Neglect Assessment Process (KF-NAP)16
* History of prior stroke
* Concurrent neurologic condition (i.e PD, TBI, MS, etc.)
* History of peripheral nerve injury
* Joint contracture or significant spasticity in the lower limbs (Modified Ashworth Scale ≥3)
* Severe knee, hip, or ankle osteoarthritis
* Severe osteoporosis as indicated by physician medical clearance
* Open wounds on surfaces in contact with exoskeleton or harness
* Unstable spine or unhealed fractures
* Weight bearing precautions
* Unresolved deep vein thrombosis (DVT)
* Concurrent participation in other lower limb research studies that according to the PI is likely to affect study outcome or confound results
* Pregnancy

EksoNR Exclusion Criteria:

* Weight >220 lbs (100 kg)
* Height below 60 inches or above 76 inches
* Standing hip width of approximately 18 inches or more
* Joint contractures or range of motion deficits that limit normal range of motion during ambulation
* Knee flexion contracture greater than 12°
* Hip flexion contracture greater than 17°
* Inability to achieve 0° neutral ankle dorsiflexion with knee flexion up to 12°
* Bilateral hip flexion less than 110°
* Leg length discrepancy
* Greater than 0.5 in. (1.27 cm) for upper legs
* Greater than 0.75 in. (1.91 cm) for lower legs
* Active heterotopic ossification
* Significant spasticity in the lower limbs (Modified Ashworth Scale ≥3)
* High anxiety or claustrophobia
* Clostridium difficile or other gastrointestinal isolation precautions
* Colostomy
* Uncontrolled autonomic dysreflexia
* Lower limb prosthesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Started | 7 | 7
Completed | 5 | 5
Not Completed | 2 | 2
Not completed — discharge to acute care prior to completion of study | 2 | 1
Not completed — patient self-withdrew from study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: The data obtained from 3 participants in each group (6 total) was analyzed due to completeness over 3 weeks.
  years | 68 [44 to 72] | 62 [53 to 72] | 65 [50.75 to 72]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The data from 3 participants in each group was analyzed due to completeness (6 total)
  Participants
    Female | 3 | 1 | 4
    Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Scale for Contraversive Pushing
Description: The Scale for Contraversive Pushing is a three-item test used to measure lateropulsion also known as contraversive pushing behaviors. It is scored on a three point ordinal scale. It rates a participant's action/reaction of maintaining or changing a position in both sitting and standing. A score >0 in each section indicates the presence of contraversive pushing behaviors. The maximum score is 6. The minimum score is 0, indicating an absence of pushing behaviors. The lower the score, the better.
Time Frame: Baseline, 3 weeks
Population: Outcome performance data was collected at baseline and at 3 weeks. Average score for each group was calculated at week 0 and week 3. The change scores from baseline to week 3 are used for this analysis. They were calculating by subtracting the average score at baseline from the average score at week 3. Due to noticeable differences in outcome performance for both groups at baseline, percent change was used to provide a more accurate comparison of changes.
Measure: Mean (Standard Deviation); unit: percent change in points
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
percent change in points | -47.01 (47.65) | -59.72 (8.67)

2. Primary Outcome: Change in Burke Lateropulsion Scale
Description: The Burke Lateropulsion Scale is a five-item test used to measure lateropulsion, scored on a four to five point ordinal scale. It rates a participant's action/reaction of keeping or changing a position in sitting, standing, rolling in supine, transfers, and walking. A lower score is better. The minimum score is 0, indicating the absence of contraversive pushing behaviors. The maximum score is 17. Research indicates a score of ≥2 as a cutoff for the presence of contraversive pushing behaviors.
Time Frame: Baseline, 3 weeks
Population: Outcome performance data was collected at baseline and at 3 weeks. Average score for each group was calculated at baseline and week 3. The change scores from baseline to week 3 are used for this analysis. They were calculated by subtracting the average score at baseline from the average score at week 3. Due to noticeable differences in outcome performance for both groups at baseline, percent change was used to provide a more accurate comparison of changes.
Measure: Mean (Standard Deviation); unit: percent change in points
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
percent change in points | -67.5 (30.31) | -53.99 (29.48)

3. Secondary Outcome: Change in 10 Meter Walk Test
Description: The 10 Meter Walk Test is a common clinical measure of gait speed. Participants are directed to walk at their comfortable, self-selected speed. Participants are positioned at the start line and instructed to walk the entire 10 meter distance while the therapist times the middle six meters. The two meter distance before and after the timed course is meant to minimize the effect of acceleration and deceleration. Time is recorded to the one hundredth of a second (example: 2.46 seconds). The test is performed two times at self-selected speed. The average of the two times is used to calculate velocity in m/s. The minimum gait speed is zero meters/second meaning the participant is unable to ambulate without someone else dependently advancing his/her limb or 2 or more people are required to assist with ambulation. There is no set maximum score. A higher score in meters/second means the participant can ambulate at a faster velocity or gait speed, which is better.
Time Frame: Baseline, 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change of velocity
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
percent change of velocity | 143.33 (176.16) | 220.37 (37.82)

4. Secondary Outcome: Change in 6 Minute Walk Test
Description: The 6 Minute Walk Test measures the distance a participant can walk indoors on a flat, hard surface in a period of six minutes. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test is self-paced. Participants are allowed to stop and rest during the test; however, the timer does not stop. If a participant is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. Appropriate assistive devices, bracing, and the minimal amount of physical assistance from the physical therapist will be applied. Minimum score is zero meters, meaning the participant is unable to ambulate in any given time. There is no set maximum score as the participant is instructed to ambulate the longest distance possible in six minutes. This test is typically measured in meters or feet. A higher value indicates the participant walked a further distance, which is better.
Time Frame: Baseline, 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in meters walked
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
percent change in meters walked | 267.65 (214.33) | 261.42 (118.97)

5. Secondary Outcome: Change in Berg Balance Scale
Description: The Berg Balance Scale is a 14-item test, scored on a five point ordinal scale. It measures functional balance in a clinical setting and includes static and dynamic tasks (such as sitting, standing, transitioning from sitting to standing, standing on one foot, retrieving an object from the floor), during which participants must maintain their balance. The minimum score is 0 and the maximum score is 56. A higher score is better.
Time Frame: Baseline, 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in points
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
percent change in points | 73.33 (88.08) | 371.67 (286.20)

6. Secondary Outcome: Change in Function in Sitting Test
Description: The Function in Sitting Test is a 14-item test of sitting balance, scored on a five point ordinal scale. It measures sensory, motor, proactive, reactive, and steady state balance factors. The minimum score is 0 and the maximum score is 56. A higher score is better.
Time Frame: Baseline, 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change in points
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
Percent change in points | 70.57 (58.68) | 58.15 (34.78)

7. Secondary Outcome: Change in Functional Independence Measure
Description: The Functional Independence Measure is an 18-item test (13 motor tasks, 5 cognitive tasks) for evaluating level of disability and how much assistance is needed for a participant to perform certain activities of daily living. Each item is scored on a seven point ordinal scale, ranging from 1point, indicating total assistance, to 7 points, indicating total independence. A higher score is better. Items include eating, grooming, bathing, dressing, toileting, bladder/bowel management, transfers, locomotion, stairs, comprehension, expression, social interaction, problem solving, and memory.
Time Frame: Baseline, 3 weeks
Population: Data was not collected for this outcome per co-investigators' decision.
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Quality Indicators
Description: This is a standardized, evidence-based measure of health care quality used to track clinical performance and outcomes in post-acute care. Items are scored on a six point ordinal scale, ranging from 6-independent to 1-dependent. A higher sore is better. Items can also be coded as participant refuses, not applicable, environmental limitations, not attempted due to medical condition or safety concerns, or unplanned discharge.
Time Frame: Baseline, 3 weeks.
Population: Data was not collected for this outcome per co-investigators' decision.
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Manual Muscle Test
Description: Manual Muscle Test is a procedure for evaluating the strength of 16 individual muscles relative to gravity and manual resistance. Instructions are provided to the participant before testing each muscle. A muscle is isolated, and gradual external force is applied at a right angle to the muscle's long axis. Each muscle is scored on a graded scale of "weak" to "strong" based on the participant's ability to resist the external force. The test is first completed for muscles on the unimpaired side to determine normal strength before being repeated on the impaired side. Weaker participants may be tested while lying prone (gravity eliminated). 0 is a minimum score and 5 is the maximum score. A higher score is better.
Time Frame: Baseline, 3 weeks
Population: This outcome measure was not collected or analyzed per investigator discretion.
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Passive Range of Motion
Description: The purpose of this test is to evaluate a participant's passive range of motion in the joints of the hips, knees, and ankles. The minimum value being 0 degrees and the maximum value varies based on joint. Normative values are different based on joint. Typically, a higher value is better.
Time Frame: Baseline, 3 weeks.
Population: Data was not collected analyzed for this outcome per co-investigators' decision. This is not typical standard of care at this inpatient of setting,
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Modified Ashworth Scale
Description: The Modified Ashworth Scale is a 6-point ordinal scale used to grade the amount of hypertonicity in individuals with neurological diagnoses. one is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner. A score of 0 (minimum) on the scale indicates no increase in tone while a score of 4 (maximum) indicates rigidity. A lower score is better.
Time Frame: Baseline, 3 weeks
Population: as for outcome 10
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Median Steps Per Session
Description: The number of steps taken during each training session will be measured using ActiGraph GT9X Link activity monitors. These devices are small accelerometers that can be worn on a belt and/or on the ankle to record steps during an activity. The therapist leading the intervention session will apply the ActiGraph at the beginning of each intervention session and remove it upon completion. The minimum number of steps is 0 and there is no maximum. A higher number of steps in considered better.
Time Frame: Week 1, Week 2, Week 3
Population: During training, the number of steps were collected for each of the three training sessions per week, over 3 weeks. The median and interquartile ranges across participants in each group was calculated for week 1, week 2 and week 3 using raw values, due to the data not being normally distributed. These values were compared between groups.
Measure: Median (Inter-Quartile Range); unit: Steps Per session
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
Steps Per session
  Week 1 Steps | 1449 [735 to 1583] | 649 [473 to 708]
  Week 2 Steps | 1513 [1353 to 2123] | 727 [725 to 891]
  Week 3 Steps | 1505 [775 to 2081] | 1091 [1074 to 1097]

13. Secondary Outcome: Maximum Heart Rate
Description: The target range of 70-85% of age-predicted maximum heart rate will be calculated for each participant utilizing HRmax = 208 - [0.7 × age] as developed by Tanaka et al in 2001. It is recommended that clinicians should apply moderate to high-intensity walking training to improve walking speed and endurance individuals poststroke. We will record the maximum heart rate, in beats per minute, achieved for participants each gait training session utilizing the Polar OH1 Optical Heart Rate Sensor. There is no maximum or minimum value for this measure. Typically, higher is better.
Time Frame: Week 1, Week 2, Week 3
Population: During training, maximum heart rate achieved was collected for participants in each of the three training sessions per week, over 3 weeks. The median and interquartile ranges for week 1, week 2 and week 3 in each group were calculated using raw values, due to the data not being normally distributed. These values were compared between groups.
Measure: Median (Inter-Quartile Range); unit: Beats per minute
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
Beats per minute
  Week 1 Maximum Heart Rate | 104 [101 to 120] | 119 [101 to 135]
  Week 2 Maximum Heart Rate | 118 [93 to 119] | 124 [109 to 132]
  Week 3 Maximum Heart rate | 118 [95 to 130] | 124 [112 to 136]

14. Secondary Outcome: Maximum Borg Rating of Perceived Exertion
Description: The Borg Rating of Perceived Exertion (RPE) is a tool to measure the subjective report of effort, exertion, and fatigue during physical work. It consists of a 15-point scale from 6-20, in which 6=no exertion and 20=absolute maximum exertion. A higher is correlated with higher intensity. It is presented to the participant in written format with descriptors to standardize the report of perceived exertion across tasks.
Time Frame: Week 1, Week 2, Week 3
Population: Maximum rate of perceived exertion (RPE) achieved was collected for participants in each of the three training sessions per week, over 3 weeks. The median and interquartile ranges for week 1, week 2 and week 3 in each group were calculated using raw values, due to the data not being normally distributed. These values were compared between groups.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 3 | 3
Score on a scale
  Week 1 Maximum RPE | 15 [14 to 15] | 14 [13 to 15]
  Week 2 Maximum RPE | 15 [15 to 16] | 16 [15 to 16]
  Week 3 Maximum RPE | 15 [14 to 17] | 14 [14 to 17]

15. Secondary Outcome: Numerical Rating Pain Scale
Description: The Numerical Rating Pain Scale is used to measure the subjective report of pain intensity. It consists of an 11-point scale, 0-10, in which zero indicates no pain and ten indicates the most intense pain imaginable. A lower sore is better.
Time Frame: Week 1, Week 2, Week 3
Population: Numeric Pain rating scale was not collected for participants per co-investigator discretion.
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 1 year period, throughout the completion of the study.
Description: All definitions are the same as described in clinicaltrials.gov definitions.
Arm/Group | Body-weight-supported Treadmill Training | EksoNR Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT04550039/Prot_002.pdf
  • Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT04550039/ICF_001.pdf